CLINICAL TRIAL: NCT02233296
Title: A Randomized Open Label Study to Compare the Bioavailability of Lasmiditan 200 mg Under Fed and Fasted Conditions in Healthy Male and Female Subjects
Brief Title: Food-Effect Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16905; H8H-CD-LAHR (Other: Eli Lilly and Company); COL MIG-104 (Other: CoLucid Pharmaceuticals)
Record Dates: First submitted 2014-08-28; First posted 2014-09-08 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Dosing Sequence: Administration of lasmiditan 200 mg in fed state in Dosing Period 1 followed by administration of lasmiditan 200 mg in fasted state in Dosing Period 2
  Interventions: Drug: Lasmiditan
- Group B (Experimental): Dosing Sequence: Administration of lasmiditan 200 mg in fasted state in Dosing Period 1 followed by administration in lasmiditan 200 mg fed state in Dosing Period 2.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — 2 discrete doses separated by 6 days.
  Other Names: COL-144; LY573144

SUMMARY:
This study will evaluate the effect of food on the pharmacokinetics (PK) of a single dose of lasmiditan in healthy participants.

DETAILED DESCRIPTION:
An open-label, cross-over, two-period, randomized, sequential study in order to investigate the effect of food on the pharmacokinetics of lasmiditan 200 mg. Two single doses of lasmiditan will be administered with the participants in fed and fasted states.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-50 years.
* Able and willing to give written informed consent.
* Females of child bearing potential must be using or willing to use a medically acceptable method (as defined by the Investigator) of birth control.
* Body mass index (BMI) within 19 and 29.9 kilograms per meter squared (kg/m²).
* No clinically significant abnormalities (as determined by the Principal Investigator) in hematology, blood chemistry and urinalysis lab tests at screening.
* No history of alcohol or drug abuse within the past year. Negative urinary drugs of abuse and alcohol screen determined within 21 days of the start of the study and at check-in Day -1.
* Must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.

Exclusion Criteria:

* Any medical condition or clinical laboratory test which in the judgment of the Investigator makes the participant unsuitable for the study.
* Pregnant or breast-feeding women.
* Use of any prescription within 14 days prior to dosing (except hormonal contraceptives) or over the-counter medications, including vitamins and herbal or dietary supplements within 7 days prior to dosing unless approved by the Investigator and Medical Monitor.
* History within the previous 3 years or current evidence of abuse of any drug, prescription or illicit, or alcohol; a positive urine screen for drugs of abuse or alcohol.
* History of orthostatic hypotension with or without syncope.
* At imminent risk of suicide (positive response to question 4 or 5 on the Columbia-Suicide Severity Rating Scale [C-SSRS]) or had a suicide attempt within 6 months prior to screening.
* Participation in any clinical trial of an experimental drug or device in the previous 30 days.
* Positive Hepatitis C antibody, Hepatitis B surface antigen, or positive human immunodeficiency virus (HIV) antibody.
* Donated plasma in the 7 days or blood in the 3 months preceding study drug administration.
* Inability to communicate well with the Investigator and study staff (i.e., language problem, poor mental development or impaired cerebral function).
* Inability to fast or consume the food provided in the study.
* Relatives of, or staff directly reporting to, the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty one (51) healthy participants were recruited according to the procedures of the Phase 1 unit. Thirty four were determined to be eligible. Thirty participants entered and completed the study.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: healthy male and female participants aged 18-
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics - Cmax (ng/mL)
Description: This study was designed to estimate the relative bioavailability of lasmiditan 200 mg in the fed state relative to the fasted state. For each primary pharmacokinetic endpoint, i.e., Area under concentration curve (time zero to last, time zero to infinity), Maximum concentration, point estimates and corresponding 90% confidence intervals were constructed. Duration of the study was approximately 5 weeks, including up to 3 weeks for screening and 16 days on study (2 - 3 day dosing periods, 6 day washout period and follow-up).
Time Frame: Sequential timepoints on each dosing day pre-dose to 30 h (timepoints - pre-dose and then 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 30 hours post dose)
Population: all participants with evaluable PK data according to the following criteria:
  * completion of both treatment regimens,
  * availability of measurements of the primary PK variable(s) for both treatments (Cmax and AUC0-inf or AUC0-t),
  * absence of any important protocol deviation that would have rendered the data incomparable between treatments
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fed Condition; Fasted Condition: Participants were randomized to dosing sequence of fed/fasted or fasted/fed. Data from specific condition (fed or fasted) were pooled for PK analysis.
Arm/Group | Fed Condition | Fasted Condition
Number analyzed (Participants) | 30 | 30
ng/mL | 394.7 (168.7) | 322.8 (122.0)

2. Primary Outcome: Pharmacokinetics - Tmax (Hours)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fed Condition | Fasted Condition
Number analyzed (Participants) | 30 | 30
hours | 2.5 (1.0) | 1.5 (1.0)

3. Secondary Outcome: Safety. Safety Measurements Include Physical Exams, Vital Signs, ECGs, Clinical Laboratory Assessments, AEs, Columbia Suicide Severity Rating Scale (C-SSRS).
Description: Safety was evaluated in all participants (n=30) under the fasted condition and the fed condition, not by sequence of assigned cross-over (fed/fasted or fasted/fed). The number of unique subjects with an AE and the number of events are provided.
Time Frame: Duration of study- From Screening (signing informed consent form) to End-of-Study ~ 15 days
Population: All the participants included in the study who received at least one dose of lasmiditan (n=30). Adverse events were considered in all participants under the fed condition and then in all participants under the fasted condition not per sequence of dosing (fed/fasted or fasted/fed).
Measure: Number; unit: participants with adverse events
Groups:
- Fed Condition: Data presented is all participants in the fed condition not by sequence of assigned cross-over (fed/fasted or fasted/fed).
- Fasted Condition: Data presented is all participants in the fasted condition, not by sequence of assigned cross-over (fed/fasted or fasted/fed).
Arm/Group | Fed Condition | Fasted Condition
Number analyzed (Participants) | 30 | 30
participants with adverse events | 19 | 23

4. Secondary Outcome: Tolerability
Description: Tolerability was defined as the number of participants that did not withdraw from the study early due to adverse events.
Time Frame: 15 days
Population: All the participants included in the study who received at least one dose of lasmiditan (n=30). Participant disposition was considered for all participants under the fed condition and then all participants under the fasted condition not per sequence of dosing (fed/fasted or fasted/fed).
Measure: Number; unit: participants
Groups:
- Fed Condition (n=30): Data presented is all participants in the fed condition, not by sequence of assigned cross-over (fed/fasted or fasted/fed).
- Fasted Condition (n=30): Data presented is all participants in the fasted condition, not by sequence of assigned cross-over (fed/fasted or fasted/fed).
Arm/Group | Fed Condition (n=30) | Fasted Condition (n=30)
Number analyzed (Participants) | 30 | 30
participants
  early withdrawals | 0 | 0
  completers | 30 | 30

5. Primary Outcome: Pharmacokinetics - AUC0-t (ng.h/mL)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: all participantss with evaluable PK data according to the following criteria:
  * completion of both treatment regimens,
  * availability of measurements of the primary PK variable(s) for both treatments (Cmax and AUC0-inf or AUC0-t),
  * absence of any important protocol deviation that would have rendered the data incomparable between treatments
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Fed Condition | Fasted Condition
Number analyzed (Participants) | 30 | 30
ng.h/mL | 2244 (926.2) | 1892 (746)

6. Primary Outcome: Pharmacokinetics - AUC0-inf (ng.h/mL)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Fed Condition | Fasted Condition
Number analyzed (Participants) | 30 | 30
ng.h/mL | 2265 (938.1) | 1906 (751.4)

ADVERSE EVENTS:
Time Frame: From signing informed consent form (ICF) to End-of-study Visit (15 days).
Description: AEs are collected from ICF until the completion of EoS/Visit 4. AEs reported prior to dosing were captured and considered non TEAEs. AEs reported more than 48 hours after dosing during the days between Dosing Period 1 and Dosing Period 2 and until the completion of EoS/Visit 4 will be captured and considered non TEAEs.
Groups:
- Fed Condition (n=30): Participants were randomized to fed/fasted or fasted/fed. Conditions were pooled for analysis so regardless of sequence all AEs reported while participant was in fed condition are considered equally.
- Fasted Condition (n=30): Participants were randomized to fed/fasted or fasted/fed. Conditions were pooled for analysis so regardless of sequence all AEs reported while participant was in fasted condition are considered equally.
Arm/Group | Fed Condition (n=30) | Fasted Condition (n=30)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 19/30 | 23/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fed Condition (n=30) (N=30) | Fasted Condition (n=30) (N=30)
ALL (Eye disorders) | 1 (1) | 0 (0)
vision blurred (Eye disorders) | 1 (1) | 0 (0)
ALL (Nervous system disorders) | 18 (24) | 23 (26)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Dizziness - Postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 18 (18) | 20 (20)
ALL (Vascular disorders) | 2 (2) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less